CLINICAL TRIAL: NCT03533608
Title: Pilot Study of Group Prolonged Exposure in Residential Treatment (CDA 15-251)
Brief Title: Optimizing Treatment Response in VA Specialized Intensive/Inpatient PTSD Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDX 18-002; CDA 15-251 (Other Grant/Funding Number: Dept of Veterans Affairs HSRD)
Record Dates: First submitted 2018-05-10; First posted 2018-05-23 (Actual); Results first posted 2021-03-05 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: PTSD
Keywords: PTSD; Prolonged Exposure; Group Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Participants will engage in 12, 90-minute sessions of Group PE over the course of 6 weeks. Treatment consists of psychoeducation, rationale for treatment, and in vivo exposure to reduce trauma-related avoidance and thereby improve PTSD symptoms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Group PE (Experimental): Participants will engage in twelve 90-minute sessions of Group PE over the course of 6 weeks. Treatment consists of psychoeducation, rationale for treatment, and in vivo exposure to reduce trauma-related avoidance and thereby improve PTSD symptoms.
  Interventions: Behavioral: Group PE

INTERVENTIONS:
Behavioral: Group PE — Participants will engage in twelve 90-minute sessions of Group PE over the course of 6 weeks. Treatment consists of psychoeducation, rationale for treatment, and in vivo exposure to reduce trauma-related avoidance and thereby improve PTSD symptoms.

SUMMARY:
Prolonged Exposure therapy (PE) is a first-line treatment for posttraumatic stress disorder; however few VA patients receive this treatment. One of the barriers to PE receipt is that this treatment is only available in an individual (one-on-one) format, whereas many VA mental health clinics provide the majority of their psychotherapy services in group format. In particular, PTSD residential rehabilitation programs (RRTPs) offer most programming in group format. Thus, the current study was designed to pilot test a group format of PE in RRTPs.

DETAILED DESCRIPTION:
Fifty Veterans who are currently receiving treatment in the PTSD RRTP at a Midwest VA will be recruited to participate in a Group PE protocol. Participants will engage in 12, 90-minute sessions of Group PE over the course of 6 weeks. Treatment consists of psychoeducation, rationale for treatment, and in vivo exposure to reduce trauma-related avoidance and thereby improve PTSD symptoms. PTSD symptoms will be measured via the PCL-5. The goal of this pilot study will be to determine whether or not it will be feasible to conduct a full-scale trial of Group PE in the current setting by testing the process, resources, management, and scientific basis of the planned trial. As such, the proposed study will primarily assess feasibility outcomes and not efficacy outcomes. The investigators will assess number of participants screened, number meeting inclusion criteria, adherence of participants to the proposed treatment (measured via number of sessions attended), standard deviation of the outcome measure (PCL-5), response rates to questionnaires, and loss to follow-up. The investigators will also measure clinicians' adherence to protocol and acceptability of the treatment to patients.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria are current engagement in treatment at the Battle Creek VA PTSD Residential Rehabilitation Treatment Program.

Exclusion Criteria:

* Exclusion criteria are severe cognitive impairment that in the judgment of the PI or the patient's clinical providers make it unlikely that the patient can adhere to the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Kaufman Sripada, PhD MS, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (2):
- United States (2):
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - Battle Creek VA Medical Center, Battle Creek, MI, Battle Creek, Michigan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group PE
Started | 39
Completed | 34
Not Completed | 5
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Population: Intent to treat analyses were performed on the 39 enrolled participants, including the 5 who left treatment early but agreed to complete follow-up assessments.
Arm/Group | Group PE
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.08 (8.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 34
  Black | 3
  Unknown | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in PTSD Symptoms
Description: PTSD symptoms will be measured via the PCL-5 at baseline, 6-week, and 2-months. The PCL-5 is a 20-item self-report measure that assesses the presence and severity of PTSD symptoms. Patients are asked to rate how bothered they are by each item in the past month on a 5-point likert scale ranging from 0-4 (not at all, a little bit, moderately, quite a bit, extremely). Items are summed together and a PCL-5 cut point score of 33 is used for provisional PTSD diagnosis. Change = (Week 6 score-Baseline score) and (2 month score-Baseline score).
Time Frame: Baseline, 6-week, and 2-months
Population: Scores are reported for the 39 enrolled participants, including the 5 who did not complete the treatment but agreed to complete the follow-up assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group PE
Number analyzed (Participants) | 39
score on a scale
  Change in Baseline to 6-weeks | -23.86 (13.81)
  Change in Baseline to 2-months | -19.51 (13.81)
Statistical Analysis 1: Comparison: Group PE; Test type: Other — Descriptive; Mean Difference (Final Values) = 19.51

2. Primary Outcome: Change in Depression Symptoms
Description: Depressive symptoms will be measured via the PHQ-9 at baseline, 6-weeks, and 2-months. The PHQ-9 is a 9-item self-report measure that assesses the presence and severity of depressive symptoms. Patients are asked to rate the presence of symptoms over the past 2 weeks on a 4-point likert scale ranging from 0-3 (not at all, several days, more than half the days, nearly every day). Individual items are summed together and Total scores ranging from 5-9 indicate mild depression, 10-14 indicate moderate depression, 15-19 indicate moderately severe depression, and 20-27 indicate severe depression. Change = (Week 6 score-Baseline score) and (2 month score-Baseline score).
Time Frame: Baseline, 6 weeks, 2-months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group PE
Number analyzed (Participants) | 39
score on a scale
  Change from baseline to 6-weeks | -4.68 (4.51)
  Change from baseline to 2-months | -4.04 (4.51)
Statistical Analysis 1: Comparison: Group PE; Test type: Other — Descriptive; Mean Difference (Final Values) = 4.04

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the participant's study involvement, which was approximately 3 months.
Arm/Group | Group PE
All-Cause Mortality (participants affected / at risk) | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-12): https://cdn.clinicaltrials.gov/large-docs/08/NCT03533608/Prot_SAP_001.pdf